CLINICAL TRIAL: NCT01964716
Title: A Phase 3, Randomized, Open-label Trial To Evaluate The Safety, Tolerability And Immunogenicity Of 13-valent Pneumococcal Conjugate Vaccine Formulated In Multidose Vials Given With Routine Pediatric Vaccinations In Healthy Infants
Brief Title: 13vPnC Multidose Vial Safety, Tolerability and Immunogenicity Study in Healthy Infants.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B4671001; 2012-000482-21 (EudraCT Number)
Record Dates: First submitted 2013-09-09; First posted 2013-10-17 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-02

CONDITIONS: Pneumococcal Vaccines
Keywords: Prevenar 13; 13vPnC; Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multidose Vial Group (Experimental): Subjects will receive three doses of 13-valent pneumococcal conjugate vaccine in the multidose vial formulation. Each dose is 0.5 mL
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine
- Single-Dose Syringe Group (Active Comparator): Subjects will receive three doses of 13-valent pneumococcal conjugate vaccine in the single-dose syringe formulation. Each dose is 0.5 mL
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — Subjects will receive three doses (0.5 mL each) of 13-valent pneumococcal conjugate vaccine (multidose vial formulation) in the anterolateral thigh muscle of the left leg. Dose 1 is administered between 42 and 70 days of age, dose 2 is administered 28 to 42 days after dose 1, dose 3 is administered 28 to 42 days after dose 2.
  Arms: Multidose Vial Group
Biological: 13-valent pneumococcal conjugate vaccine — Subjects will receive three doses (0.5 mL each) of 13-valent pneumococcal conjugate vaccine (single-dose syringe formulation) in the anterolateral thigh muscle of the left leg. Dose 1 is administered between 42 and 70 days of age, dose 2 is administered 28 to 42 days after dose 1, dose 3 is administered 28 to 42 days after dose 2.
  Arms: Single-Dose Syringe Group

SUMMARY:
This study will compare the immune responses of the infants who have been given 13vPnC in the mutidose vial formulation to the immune reponses of the infants who have been given 13vPnC in the single-dose syringe formulation.

It will also evaluate the safety of 13-valent pneumococcal conjugate vaccine (13vPnC) in all infants who are vaccinated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 42 to 70 days at enrollment.
* Determined by medical history, physical examination, and clinical judgment to be eligible for the study
* Weight of 3.5 kg or greater at the time of enrollment

Exclusion Criteria:

* Previous vaccination with licensed or investigational pneumococcal vaccine.
* A previous anaphylactic reaction to any vaccine or vaccine-related component.
* Contraindication to vaccination with pneumococcal conjugate vaccine.
* Receipt of blood products or gamma-globulin since birth

Ages: 42 Days to 70 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- The Gambia (2):
  - Medical Research Council Unit, The Gambia, Fajara, The Gambia, West Africa
  - Fajikunda Major Health Centre, Ksmd, The Gambia

REFERENCES:
- [Derived] Idoko OT, Mboizi RB, Okoye M, Laudat F, Ceesay B, Liang JZ, Le Dren-Narayanin N, Jansen KU, Gurtman A, Center KJ, Scott DA, Kampmann B, Roca A. Immunogenicity and safety of 13-valent pneumococcal conjugate vaccine (PCV13) formulated with 2-phenoxyethanol in multidose vials given with routine vaccination in healthy infants: An open-label randomized controlled trial. Vaccine. 2017 May 31;35(24):3256-3263. doi: 10.1016/j.vaccine.2017.04.049. Epub 2017 May 4. PMID 28479175
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4671001&StudyName=13vPnC%20Multidose%20Vial%20Safety%2C%20Tolerability%20and%20Immunogenicity%20Study%20in%20Healthy%20Infants.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total number of participants screened were 526, out of which 500 were enrolled in the study. The study was conducted in Gambia which started on 09 January 2014 and completed on 01 September 2014.
Groups:
- 13vPnC Multi-dose Vial (MDV): Participants received three doses of 0.5 milliliter (mL) of 13-valent pneumococcal conjugate vaccine (13vPnC) with 2-phenoxyethanol (2-PE) in MDV intramuscularly at 8, 12 and 16 weeks of age.
- 13vPnC Single-Dose Syringe (SDS): Participants received three doses of 0.5 milliliter (mL) of 13-valent pneumococcal conjugate vaccine (13vPnC) without 2-phenoxyethanol (2-PE) in SDS intramuscularly at 8, 12 and 16 weeks of age.
Period: Overall Study
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS)
Started | 250 | 250
Vaccinated Dose 1 | 250 | 250
Vaccinated Dose 2 | 249 | 248
Vaccinated Dose 3 | 247 | 244
Completed | 245 | 244
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — No longer met eligibility criteria | 1 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS) | Total
Number analyzed (Participants) | 250 | 250 | 500
Age, Continuous [Mean (Standard Deviation); unit: days] | 57.3 (8.6) | 56.9 (8.8) | 57.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 130 | 259
  Male | 121 | 120 | 241

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Antibody Concentration Greater Than or Equal To (>=) 0.35 Microgram Per Milliliter (mcg/mL) 1 Month After the Infant Series for Each Vaccine Group
Description: Percentage of participants achieving predefined antibody threshold >=0.35 mcg/mL along with the corresponding 95% confidence interval (CI) for the 13 pneumococcal serotypes (serotypes 1, 3, 4, 5, 6A, 6B, 7F 9V, 14, 18C, 19A, 19F and 23F) are presented. Exact 2-sided confidence interval (Clopper and Pearson) based on the observed proportion of participants. Here "n"= participants with valid and determinate IgG concentration to the given serotype.
Time Frame: 1 month after the infant series
Population: Evaluable immunogenicity population: eligible participants who received vaccine (as randomized) at all 3 doses, had blood drawn within protocol-specified time frames, had at least 1 valid and determinate assay result for proposed analysis, had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS)
Number analyzed (Participants) | 245 | 244
percentage of participants
  Serotype 1 (n=245,244) | 99.2 [97.1 to 99.9] | 100.0 [98.5 to 100.0]
  Serotype 3 (n=245,243) | 98.8 [96.5 to 99.7] | 99.6 [97.7 to 100.0]
  Serotype 4 (n=245,244) | 99.6 [97.7 to 100.0] | 99.6 [97.7 to 100.0]
  Serotype 5 (n=245,244) | 95.9 [92.6 to 98.0] | 97.1 [94.2 to 98.8]
  Serotype 6A (n=243,244) | 96.3 [93.1 to 98.3] | 97.5 [94.7 to 99.1]
  Serotype 6B (n=245,244) | 95.1 [91.6 to 97.4] | 95.1 [91.6 to 97.4]
  Serotype 7F (n=245,244) | 99.6 [97.7 to 100.0] | 100.0 [98.5 to 100.0]
  Serotype 9V (n=245,244) | 98.0 [95.3 to 99.3] | 98.4 [95.9 to 99.6]
  Serotype 14 (n=245,244) | 97.6 [94.7 to 99.1] | 98.4 [95.9 to 99.6]
  Serotype 18C (n=245,244) | 99.2 [97.1 to 99.9] | 98.0 [95.3 to 99.3]
  Serotype 19A (n=245,244) | 99.6 [97.7 to 100.0] | 98.8 [96.4 to 99.7]
  Serotype 19F (n=245,244) | 96.7 [93.7 to 98.6] | 97.1 [94.2 to 98.8]
  Serotype 23F (n=245,244) | 95.9 [92.6 to 98.0] | 95.9 [92.6 to 98.0]
Statistical Analysis 1: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 1: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC MDV - 13vPnC SDS, expressed as a percentage was analyzed; Test type: Non-Inferiority or Equivalence — Non-inferiority for a given antibody was demonstrated if the lower bound of the 2-sided, 97.5% confidence interval, computed using the Chan and Zhang procedure, for the difference in proportions (13vPnC MDV - 13vPnC SDS) was greater than -0.10; percent difference = -0.8, 97.5% CI 2-sided [-3.4 to 1.2]
Statistical Analysis 2: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 3: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC MDV - 13vPnC SDS, expressed as a percentage was analyzed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; percent difference = -0.8, 97.5% CI 2-sided [-3.7 to 1.6]
Statistical Analysis 3: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 4: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC MDV - 13vPnC SDS, expressed as a percentage was analyzed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; percent difference = 0.0, 97.5% CI 2-sided [-2.3 to 2.4]
Statistical Analysis 4: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 5: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC MDV - 13vPnC SDS, expressed as a percentage was analyzed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; percent difference = -1.2, 97.5% CI 2-sided [-5.4 to 2.8]
Statistical Analysis 5: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 6A: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC MDV - 13vPnC SDS, expressed as a percentage was analyzed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; percent difference = -1.2, 97.5% CI 2-sided [-5.3 to 2.6]
Statistical Analysis 6: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 6B: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC MDV - 13vPnC SDS, expressed as a percentage was analyzed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; percent difference = 0.0, 97.5% CI 2-sided [-4.7 to 4.7]
Statistical Analysis 7: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 7F: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC MDV - 13vPnC SDS, expressed as a percentage was analyzed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; percent difference = -0.4, 97.5% CI 2-sided [-2.7 to 1.6]
Statistical Analysis 8: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 9V: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC MDV - 13vPnC SDS, expressed as a percentage was analyzed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; percent difference = -0.4, 97.5% CI 2-sided [-3.8 to 2.8]
Statistical Analysis 9: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 14: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC MDV - 13vPnC SDS, expressed as a percentage was analyzed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; percent difference = -0.8, 97.5% CI 2-sided [-4.3 to 2.5]
Statistical Analysis 10: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 18C: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC MDV - 13vPnC SDS, expressed as a percentage was analyzed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; percent difference = 1.2, 97.5% CI 2-sided [-1.6 to 4.5]
Statistical Analysis 11: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 19A: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC MDV - 13vPnC SDS, expressed as a percentage was analyzed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; percent difference = 0.8, 97.5% CI 2-sided [-1.6 to 3.6]
Statistical Analysis 12: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 19F: Exact 2-sided confidence interval (based on Chan & Zhang) for the difference in proportions, 13vPnC multidose vial (MDV) - 13vPnC single-dose syringe (SDS), expressed as a percentage was analyzed; Test type: Superiority or Other; percentage difference = -0.4, 97.5% CI 2-sided [-4.4 to 3.5]
Statistical Analysis 13: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 23F: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC MDV - 13vPnC SDS, expressed as a percentage was analyzed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; percent difference = 0.0, 97.5% CI 2-sided [-4.3 to 4.4]

2. Primary Outcome: Geometric Mean Concentration (GMC) for Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After the Infant Series for Each Vaccine Group
Description: Antibody GMC for the 13 pneumococcal serotypes (serotypes 1, 3, 4, 5, 6A, 6B, 7F 9V, 14, 18C, 19A, 19F and 23F) are presented. GMC (13vPnC) and corresponding 2-sided 95% CI were evaluated. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw. CIs were back transformations of a confidence interval based on the Student t distribution for the mean logarithm of the concentrations. Here "n"= participants with valid and determinate IgG concentration to the given serotype.
Time Frame: 1 month after the infant series
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (mcg/mL)
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS)
Number analyzed (Participants) | 245 | 244
microgram per milliliter (mcg/mL)
  Serotype 1 (n=245,244) | 4.59 [4.11 to 5.12] | 4.45 [4.01 to 4.93]
  Serotype 3 (n=245,243) | 1.38 [1.29 to 1.49] | 1.74 [1.62 to 1.87]
  Serotype 4 (n=245,244) | 5.30 [4.84 to 5.81] | 5.28 [4.76 to 5.85]
  Serotype 5 (n=245,244) | 2.00 [1.79 to 2.22] | 1.98 [1.79 to 2.20]
  Serotype 6A (n=243,244) | 2.25 [2.02 to 2.50] | 2.19 [1.96 to 2.44]
  Serotype 6B (n=245,244) | 3.42 [2.91 to 4.02] | 3.24 [2.77 to 3.78]
  Serotype 7F (n=245,244) | 3.92 [3.59 to 4.27] | 4.18 [3.83 to 4.55]
  Serotype 9V (n=245,244) | 2.83 [2.56 to 3.13] | 2.75 [2.49 to 3.04]
  Serotype 14 (n=245,244) | 4.78 [4.06 to 5.63] | 4.96 [4.27 to 5.77]
  Serotype 18C (n=245,244) | 3.47 [3.17 to 3.79] | 2.72 [2.46 to 3.00]
  Serotype 19A (n=245,244) | 6.49 [5.70 to 7.38] | 6.44 [5.66 to 7.32]
  Serotype 19F (n=245,244) | 5.19 [4.59 to 5.86] | 5.00 [4.43 to 5.63]
  Serotype 23F (n=245,244) | 2.61 [2.30 to 2.97] | 2.17 [1.92 to 2.46]
Statistical Analysis 1: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 1: Ratio of GMCs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale; CIs for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Non-Inferiority or Equivalence — Non-inferiority for a given antibody serotype was declared if lower bound of the 2-sided, 97.5% confidence interval for the geometric mean concentration ratio (GMC MDV /GMC SDS) was greater than 0.5 (2-fold criterion); GMC Ratio = 1.03, 97.5% CI 2-sided [0.87 to 1.22]
Statistical Analysis 2: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 3: Ratio of GMCs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale; CIs for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMC Ratio = 0.79, 97.5% CI 2-sided [0.71 to 0.90]
Statistical Analysis 3: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 4: Ratio of GMCs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale; CIs for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMC Ratio = 1.00, 97.5% CI 2-sided [0.86 to 1.18]
Statistical Analysis 4: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 5: Ratio of GMCs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale; CIs for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMC Ratio = 1.01, 97.5% CI 2-sided [0.85 to 1.19]
Statistical Analysis 5: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 6A: Ratio of GMCs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale; CIs for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMC Ratio = 1.03, 97.5% CI 2-sided [0.86 to 1.22]
Statistical Analysis 6: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 6B: Ratio of GMCs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale; CIs for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMC Ratio = 1.06, 97.5% CI 2-sided [0.82 to 1.36]
Statistical Analysis 7: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 7F: Ratio of GMCs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale; CIs for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMC Ratio = 0.94, 97.5% CI 2-sided [0.82 to 1.08]
Statistical Analysis 8: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 9V: Ratio of GMCs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale; CIs for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMC Ratio = 1.03, 97.5% CI 2-sided [0.87 to 1.21]
Statistical Analysis 9: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 14: Ratio of GMCs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale; CIs for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMC Ratio = 0.96, 97.5% CI 2-sided [0.75 to 1.24]
Statistical Analysis 10: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 18C: Ratio of GMCs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale; CIs for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMC Ratio = 1.28, 97.5% CI 2-sided [1.09 to 1.49]
Statistical Analysis 11: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 19A: Ratio of GMCs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale; CIs for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMC Ratio = 1.01, 97.5% CI 2-sided [0.82 to 1.24]
Statistical Analysis 12: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 19F: Ratio of GMCs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale; CIs for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMC Ratio = 1.04, 97.5% CI 2-sided [0.85 to 1.26]
Statistical Analysis 13: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 23F: Ratio of GMCs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale; CIs for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMC Ratio = 1.20, 97.5% CI 2-sided [0.98 to 1.48]

3. Primary Outcome: Number of Participants Reporting Local Reaction Within 5 Days After Dose 1 in MDV and SDS Group
Description: Local reactions were reported within 5 days (day 2 to day 6) using an electronic diary. Tenderness was scaled as Any (tenderness present); Mild (hurt if gently touched; Moderate (hurt if gently touched with crying); Severe (caused limitation of limb movement). Redness and swelling were scaled as Any (redness or swelling present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.1 to 7.0 cm); Severe (greater than [>] 7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 5 days after Dose 1(Day 2 to Day 6) of the infant series
Population: Safety population included participants who received at least 1 dose of study vaccine. 'N' (number of participants analyzed) included participants whose response was "Yes" for any day or "No" for all days.
Measure: Number; unit: participants
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS)
Number analyzed (Participants) | 248 | 250
participants
  Redness: Any | 1 | 0
  Redness: Mild | 1 | 0
  Redness: Moderate | 0 | 0
  Redness: Severe | 0 | 0
  Swelling: Any | 1 | 0
  Swelling: Mild | 1 | 0
  Swelling: Moderate | 0 | 0
  Swelling: Severe | 0 | 0
  Tenderness: Any | 42 | 47
  Tenderness: Mild | 32 | 37
  Tenderness: Moderate | 13 | 14
  Tenderness: Severe | 0 | 0

4. Primary Outcome: Number of Participants Reporting Local Reaction Within 5 Days After Dose 2 in MDV and SDS Group
Description: as for outcome 3
Time Frame: Within 5 days after Dose 2 (Day 2 to Day 6) of the infant series
Population: Safety population included participants who received at least 1 dose of study vaccine. 'N' (number of participants analyzed) included participants whose response was "Yes" for any day or "No" for all days and 'n' = participants whose response was "Yes" for any day or "No" for all days for specified local reaction.
Measure: Number; unit: participants
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS)
Number analyzed (Participants) | 248 | 247
participants
  Redness: Any (n=247, 247) | 2 | 0
  Redness: Mild (n=247, 247) | 2 | 0
  Redness: Moderate (n=247, 247) | 0 | 0
  Redness: Severe (n=247, 247) | 0 | 0
  Swelling: Any (n=247, 247) | 2 | 0
  Swelling: Mild (n=247, 247) | 2 | 0
  Swelling: Moderate (n=247, 247) | 1 | 0
  Swelling: Severe (n=247, 247) | 0 | 0
  Tenderness: Any (n=248, 247) | 34 | 32
  Tenderness: Mild (n=248, 247) | 27 | 28
  Tenderness: Moderate (n=247, 247) | 7 | 5
  Tenderness: Severe (n=247, 247) | 0 | 0

5. Primary Outcome: Number of Participants Reporting Local Reaction Within 5 Days After Dose 3 in MDV and SDS Group
Description: as for outcome 3
Time Frame: Within 5 days after Dose 3 (Day 2 to Day 6) of the infant series
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS)
Number analyzed (Participants) | 246 | 241
participants
  Redness: Any | 0 | 0
  Redness: Mild | 0 | 0
  Redness: Moderate | 0 | 0
  Redness: Severe | 0 | 0
  Swelling: Any | 0 | 0
  Swelling: Mild | 0 | 0
  Swelling: Moderate | 0 | 0
  Swelling: Severe | 0 | 0
  Tenderness: Any | 37 | 35
  Tenderness: Mild | 30 | 32
  Tenderness: Moderate | 9 | 4
  Tenderness: Severe | 0 | 0

6. Primary Outcome: Number of Participants Reporting Systemic Events Within 5 Days After Dose 1 in MDV and SDS Group
Description: Systemic events (any fever greater than or equal to [>=] 38.0 degrees Celsius [C], decreased appetite was scaled as; Moderate (decreased oral intake); Severe (refusal to feed). Irritability scaled as; Mild (easily consolable); Moderate (requiring increased attention); Severe (Inconsolable, crying that cannot be comforted). Increased sleep was scale as; mild (increased or prolonged sleeping bouts); Moderate (slightly subdued interfering with daily activity); Severe (Disabling not interested in usual daily activity) and use of antipyretic medication were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 5 days after Dose 1 (Day 2 to Day 6) of infant series
Population: Safety population included participants who received at least 1 dose of study vaccine. 'N' (number of participants analyzed) included participants whose response was "Yes" for any day or "No" for all days. 'n' included participants whose response was "Yes" for any day or "No" for all days for specified systemic event.
Measure: Number; unit: participants
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS)
Number analyzed (Participants) | 249 | 250
participants
  Fever: >=38.0 degree C (n=248, 250) | 9 | 7
  Fever: >=38.0 but <=39.0 degrees C (n=248, 250) | 9 | 7
  Fever: >39.0 but <=40.0 degrees C (n=248, 250) | 0 | 0
  Fever: >40.0 degrees C (n=248, 250) | 0 | 0
  Decreased appetite: Any (n=248, 250) | 17 | 26
  Decreased appetite: Moderate (n=248, 250) | 17 | 26
  Decreased appetite: Severe (n=248, 250) | 0 | 0
  Irritability: Any (n=249, 250) | 103 | 93
  Irritability: Mild (n=249, 250) | 86 | 77
  Irritability: Moderate (n=248, 250) | 19 | 17
  Irritability: Severe (n=248, 250) | 0 | 0
  Increased sleep: Any (n=248, 250) | 16 | 14
  Increased sleep: Mild (n=248, 250) | 11 | 10
  Increased sleep: Moderate (n=248, 250) | 6 | 4
  Increased sleep: Severe (n=248, 250) | 0 | 0
  Use of antipyretic medication (n=248, 250) | 55 | 58

7. Primary Outcome: Number of Participants Reporting Systemic Events Within 5 Days After Dose 2 in MDV and SDS Group
Description: as for outcome 6
Time Frame: Within 5 days after Dose 2 (Day 2 to Day 6) of infant series
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS)
Number analyzed (Participants) | 248 | 247
participants
  Fever: >=38.0 degree C (n=247, 247) | 7 | 7
  Fever: >=38.0 but <=39.0 degrees C (n=247, 247) | 7 | 7
  Fever: >39.0 but <=40.0 degrees C (n=247, 247) | 1 | 0
  Fever: >40.0 degrees C (n=247, 247) | 0 | 0
  Decreased appetite: Any(n=247, 247) | 28 | 18
  Decreased appetite: Moderate (n=247, 247) | 28 | 18
  Decreased appetite: Severe (n=247, 247) | 0 | 0
  Irritability: Any (n=248, 247) | 93 | 83
  Irritability: Mild (n=248, 247) | 75 | 67
  Irritability: Moderate (n=247, 247) | 23 | 17
  Irritability: Severe (n=247, 247) | 0 | 3
  Increased sleep: Any (n=247, 247) | 24 | 14
  Increased sleep: Mild (n=247, 247) | 20 | 12
  Increased sleep: Moderate (n=247, 247) | 4 | 1
  Increased sleep: Severe (n=247, 247) | 0 | 1
  Use of antipyretic medication (n=248, 247) | 46 | 43

8. Primary Outcome: Number of Participants Reporting Systemic Events Within 5 Days After Dose 3 in MDV and SDS Group
Description: as for outcome 6
Time Frame: Within 5 days after Dose 3 (Day 2 to Day 6) of infant series
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS)
Number analyzed (Participants) | 246 | 243
participants
  Fever: >=38.0 degree C (n=246, 241) | 3 | 8
  Fever: >=38.0 but <=39.0 degrees C (n=246, 241) | 3 | 7
  Fever: >39.0 but <=40.0 degrees C (n=246, 241) | 0 | 1
  Fever: >40.0 degrees C (n=246, 241) | 0 | 0
  Decreased appetite: Any (n=246, 242) | 24 | 20
  Decreased appetite: Moderate (n=246, 242) | 24 | 19
  Decreased appetite: Severe (n=246, 241) | 0 | 1
  Irritability: Any (n=246, 243) | 83 | 92
  Irritability: Mild (n=246, 242) | 71 | 74
  Irritability: Moderate (n=246, 242) | 15 | 18
  Irritability: Severe (n=246, 241) | 1 | 5
  Increased sleep: Any (n=246, 241) | 12 | 12
  Increased sleep: Mild (n=246, 241) | 10 | 11
  Increased sleep: Moderate (n=246, 241) | 2 | 1
  Increased sleep: Severe (n=246, 241) | 1 | 0
  Use of antipyretic medication (n=246, 241) | 34 | 36

9. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) in the Infant Series
Description: An AE was any untoward medical occurrence in a participants who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 to 42 days after last dose that were absent before treatment or that worsened relative to pretreatment state
Time Frame: Dose 1 up to 28 to 42 days after dose 3
Population: Safety population included all participants who received at least 1 dose of study vaccine.
Measure: Number; unit: participants
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS)
Number analyzed (Participants) | 250 | 250
participants
  AEs | 123 | 127
  SAEs | 1 | 0

10. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) Prior to Dose 1
Description: An AE was any untoward medical occurrence in a participants who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Adverse events were also reported in participants who provided consent but were not randomized in this study. The data of these participants has been reported under 'Screened Only' arm.
Time Frame: Informed consent up to Dose 1
Population: Safety population: participants who received at least 1 dose of study vaccine. Here "N"= participants evaluable for this outcome measure.
Measure: Number; unit: participants
Groups:
- Screened Only: Participants who were screened for this study but were not randomized, assessed between signing of informed consent form and before randomization.
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS) | Screened Only
Number analyzed (Participants) | 250 | 250 | 26
participants
  AEs | 2 | 0 | 9
  SAEs | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants Achieving a Serotype-Specific Opsonophagocytic Activity (OPA) Titer >= Lower Limit of Quantitation (LLOQ) 1 Month After Infant Series
Description: Percentage of participants achieving OPA Titer >= lower limit of quantitation (LLOQ) along with 95% CI for the 13 pneumococcal serotypes (serotypes 1, 3, 4, 5, 6A, 6B, 7F 9V, 14, 18C, 19A, 19F and 23F) are presented. The LLOQ in titers for each serotype was: Pn001, 18; Pn003, 12; Pn004, 21; Pn005, 29; Pn06A, 37; Pn06B, 43, Pn7F, 210; Pn09V, 345; Pn014, 35; Pn18C, 31; Pn19A, 18; Pn19F, 48; and Pn23F, 13. Exact 2-sided confidence interval (Clopper and Pearson) based on the observed proportion of participants. Here "n"= Number of participants with an antibody titer ≥ LLOQ for the given serotype.
Time Frame: 1 month after the infant series
Population: Evaluable immunogenicity population:participants who received vaccine (randomized) at all 3 doses, had blood drawn within protocol-specified time frames, had at least 1 valid and determinate assay result for proposed analysis, had no major protocol violations. OPA analysis was performed in a subset of randomly selected participants from each group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS)
Number analyzed (Participants) | 160 | 160
percentage of participants
  Serotype 1 (n=159,160) | 71.7 [64.0 to 78.5] | 79.4 [72.3 to 85.4]
  Serotype 3 (n=160,160) | 98.8 [95.6 to 99.8] | 100.0 [97.7 to 100.0]
  Serotype 4 (n=159,159) | 100.0 [97.7 to 100.0] | 100.0 [97.7 to 100.0]
  Serotype 5 (n=160,159) | 83.1 [76.4 to 88.6] | 85.5 [79.1 to 90.6]
  Serotype 6A (n=160,160) | 99.4 [96.6 to 100.0] | 99.4 [96.6 to 100.0]
  Serotype 6B (n=156,155) | 96.8 [92.7 to 99.0] | 96.8 [92.6 to 98.9]
  Serotype 7F (n=159,160) | 100.0 [97.7 to 100.0] | 100.0 [97.7 to 100.0]
  Serotype 9V (n=158,160) | 79.7 [72.6 to 85.7] | 75.0 [67.6 to 81.5]
  Serotype 14 (n=157,160) | 81.5 [74.6 to 87.3] | 89.4 [83.5 to 93.7]
  Serotype 18C (n=159,160) | 99.4 [96.5 to 100.0] | 99.4 [96.6 to 100.0]
  Serotype 19A (n=160,160) | 95.6 [91.2 to 98.2] | 97.5 [93.7 to 99.3]
  Serotype 19F (n=158,159) | 93.7 [88.7 to 96.9] | 94.3 [89.5 to 97.4]
  Serotype 23F (n=159,160) | 96.2 [92.0 to 98.6] | 97.5 [93.7 to 99.3]
Statistical Analysis 1: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; percent difference = -7.7, 95% CI 2-sided [-17.2 to 1.9]
Statistical Analysis 2: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; percent difference = -1.2, 95% CI 2-sided [-4.4 to 1.1]
Statistical Analysis 3: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; percent difference = 0.0, 95% CI 2-sided [-2.3 to 2.3]
Statistical Analysis 4: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; percent difference = -2.4, 95% CI 2-sided [-10.6 to 5.7]
Statistical Analysis 5: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; percent difference = 0.0, 95% CI 2-sided [-2.9 to 2.8]
Statistical Analysis 6: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; percent difference = 0.0, 95% CI 2-sided [-4.5 to 4.6]
Statistical Analysis 7: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; percent difference = 0.0, 95% CI 2-sided [-2.3 to 2.3]
Statistical Analysis 8: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; percent difference = 4.7, 95% CI 2-sided [-4.5 to 14.1]
Statistical Analysis 9: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; percent difference = -7.8, 95% CI 2-sided [-15.8 to -0.0]
Statistical Analysis 10: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; percent difference = -0.0, 95% CI 2-sided [-2.9 to 2.9]
Statistical Analysis 11: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; percent difference = -1.9, 95% CI 2-sided [-6.6 to 2.4]
Statistical Analysis 12: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 19F: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC MDV - 13vPnC SDS, expressed as a percentage was analyzed; Test type: Superiority or Other; percent difference = -0.7, 95% CI 2-sided [-6.3 to 4.9]
Statistical Analysis 13: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; percent difference = -1.3, 95% CI 2-sided [-5.8 to 3.0]

12. Secondary Outcome: Serotype-Specific Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) 1 Month After the Infant Series
Description: Antibody geometric mean titers as measured by OPA assay for the 13 pneumococcal serotypes (serotypes 1, 3, 4, 5, 6A, 6B, 7F 9V, 14, 18C, 19A, 19F and 23F) are presented. GMTs were calculated using all participants with available data for the specified blood draw. CIs were back transformations of a confidence interval based on the Student t distribution for the mean logarithm of the titers. Here "n"= participants evaluable =specified category.
Time Frame: 1 month after the infant series
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC Multi-dose Vial (MDV) | 13vPnC Single-Dose Syringe (SDS)
Number analyzed (Participants) | 160 | 160
titer
  Serotype 1 (n=159,160) | 48 [39.0 to 58.0] | 52 [43.2 to 62.6]
  Serotype 3 (n=160,160) | 97 [87.3 to 108.8] | 122 [110.1 to 135.7]
  Serotype 4 (n=159,159) | 1666 [1412.3 to 1966.3] | 1492 [1285.2 to 1732.3]
  Serotype 5 (n=160,159) | 79 [67.7 to 92.4] | 80 [69.1 to 92.6]
  Serotype 6A (n=160,160) | 1690 [1460.5 to 1955.9] | 1968 [1698.5 to 2279.3]
  Serotype 6B (n=156,155) | 1990 [1611.7 to 2456.9] | 2014 [1639.1 to 2475.4]
  Serotype 7F (n=159,160) | 2891 [2565.4 to 3258.5] | 3450 [3014.7 to 3947.9]
  Serotype 9V (n=158,160) | 709 [600.5 to 836.2] | 706 [597.0 to 835.3]
  Serotype 14 (n=157,160) | 567 [415.4 to 773.5] | 786 [607.8 to 1015.3]
  Serotype 18C (n=159,160) | 2792 [2387.5 to 3264.8] | 1605 [1352.0 to 1904.4]
  Serotype 19A (n=160,160) | 305 [256.2 to 362.9] | 329 [284.8 to 379.8]
  Serotype 19F (n=158,159) | 430 [357.6 to 517.1] | 470 [391.4 to 565.3]
  Serotype 23F (n=159,160) | 918 [729.0 to 1156.4] | 998 [810.6 to 1229.6]
Statistical Analysis 1: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 1: Ratio of GMTs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Superiority or Other; GMT Ratio = 0.9, 95% CI 2-sided [0.70 to 1.20]
Statistical Analysis 2: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 3: Ratio of GMTs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Superiority or Other; GMT Ratio = 0.8, 95% CI 2-sided [0.69 to 0.93]
Statistical Analysis 3: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 4: Ratio of GMTs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Superiority or Other; GMT Ratio = 1.1, 95% CI 2-sided [0.89 to 1.39]
Statistical Analysis 4: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 5: Ratio of GMTs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Superiority or Other; GMT Ratio = 1.0, 95% CI 2-sided [0.80 to 1.22]
Statistical Analysis 5: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 6A: Ratio of GMTs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Superiority or Other; GMT Ratio = 0.9, 95% CI 2-sided [0.70 to 1.06]
Statistical Analysis 6: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 6B: Ratio of GMTs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Superiority or Other; GMT Ratio = 1.0, 95% CI 2-sided [0.74 to 1.33]
Statistical Analysis 7: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 7F: Ratio of GMTs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Superiority or Other; GMT Ratio = 0.8, 95% CI 2-sided [0.70 to 1.00]
Statistical Analysis 8: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 9V: Ratio of GMTs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Superiority or Other; GMT Ratio = 1.0, 95% CI 2-sided [0.79 to 1.27]
Statistical Analysis 9: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 14: Ratio of GMTs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Superiority or Other; GMT Ratio = 0.7, 95% CI 2-sided [0.48 to 1.08]
Statistical Analysis 10: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 18C: Ratio of GMTs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Superiority or Other; GMT Ratio = 1.7, 95% CI 2-sided [1.38 to 2.19]
Statistical Analysis 11: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 19A: Ratio of GMTs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Superiority or Other; GMT Ratio = 0.9, 95% CI 2-sided [0.74 to 1.16]
Statistical Analysis 12: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 19F: Ratio of GMTs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Superiority or Other; GMT Ratio = 0.9, 95% CI 2-sided [0.71 to 1.18]
Statistical Analysis 13: Comparison: 13vPnC Multi-dose Vial (MDV) vs 13vPnC Single-Dose Syringe (SDS); Serotype 23F: Ratio of GMTs, MDV to SDS, was calculated by back transforming the mean difference between the vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC MDV - 13vPnC SDS); Test type: Superiority or Other; GMT Ratio = 0.9, 95% CI 2-sided [0.67 to 1.25]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs)/serious AEs (SAEs): recorded from signing of informed consent form to 28 to 42 days after dose 3. Pre-specified AEs were recorded in an electronic diary: local reactions, systemic events (Day 2 to Day 6 after each vaccination)
Description: SAEs, AEs grouped by system organ class and summarized. AEs included AEs collected in electronic diary (local, systemic reactions;systematic assessment), events collected on case report form at each visit (non-systematic assessment). AEs also reported in participants who provided consent but were not randomized (reported under 'Screened Only' arm).
Groups:
- 13vPnC MDV: Informed Consent to Dose 1: Participants who were randomized to receive 13vPnC (PF-06414256) MDV at 8, 12, and 16 weeks of age, assessed between signing of informed consent and before Dose 1.
- 13vPnC SDS: Informed Consent to Dose 1: Participants who were randomized to receive 13vPnC (PF-05208760) SDS at 8, 12, and 16 weeks of age, assessed between signing of informed consent and before Dose 1.
- 13vPnC MDV: After Dose 1: Participants who received single 0.5 mL dose of 13vPnC (PF-06414256) using MDV intramuscularly into the anterolateral thigh muscle of the left leg at 8 weeks of age, assessed after Dose 1 and before Dose 2.
- 13vPnC SDS: After Dose 1: Participants who received single 0.5 mL dose of 13vPnC (PF-05208760) using SDS intramuscularly into the anterolateral thigh muscle of the left leg at 8 weeks of age, assessed after Dose 1 and before Dose 2.
- 13vPnC MDV: After Dose 2: Participants who received two 0.5 mL doses of 13vPnC (PF-06414256) using MDV intramuscularly into the anterolateral thigh muscle of the left leg 8, 12 weeks of age, assessed after Dose 2 and before Dose 3.
- 13vPnC SDS: After Dose 2: Participants who received two 0.5 mL doses of 13vPnC (PF-05208760) using SDS intramuscularly into the anterolateral thigh muscle of the left leg 8, 12 weeks of age, assessed after Dose 2 and before Dose 3.
- 13vPnC MDV: After Dose 3: Participants who received all three 0.5mL doses of 13vPnC (PF-06414256) using MDV intramuscularly into the anterolateral thigh muscle of the left leg at 8 weeks of age, assessed after Dose 3 and up to blood draw at 4 weeks.
- 13vPnC SDS: After Dose 3: Participants who received all three 0.5mL doses of 13vPnC (PF-05208760) using SDS intramuscularly into the anterolateral thigh muscle of the left leg at 8 weeks of age, assessed after Dose 3 and up to blood draw at 4 weeks.
Arm/Group | 13vPnC MDV: Informed Consent to Dose 1 | 13vPnC SDS: Informed Consent to Dose 1 | 13vPnC MDV: After Dose 1 | 13vPnC SDS: After Dose 1 | 13vPnC MDV: After Dose 2 | 13vPnC SDS: After Dose 2 | 13vPnC MDV: After Dose 3 | 13vPnC SDS: After Dose 3 | Screened Only
Serious Adverse Events (participants affected / at risk) | 0/250 | 0/250 | 0/250 | 0/250 | 0/249 | 0/248 | 1/247 | 0/244 | 0/26
Other Adverse Events (participants affected / at risk) | 2/250 | 0/250 | 113/250 | 107/250 | 114/249 | 99/248 | 97/247 | 102/244 | 9/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC MDV: Informed Consent to Dose 1 (N=250) | 13vPnC SDS: Informed Consent to Dose 1 (N=250) | 13vPnC MDV: After Dose 1 (N=250) | 13vPnC SDS: After Dose 1 (N=250) | 13vPnC MDV: After Dose 2 (N=249) | 13vPnC SDS: After Dose 2 (N=248) | 13vPnC MDV: After Dose 3 (N=247) | 13vPnC SDS: After Dose 3 (N=244) | Screened Only (N=26)
Sudden infant death syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 13vPnC MDV: Informed Consent to Dose 1 (N=250) | 13vPnC SDS: Informed Consent to Dose 1 (N=250) | 13vPnC MDV: After Dose 1 (N=250) | 13vPnC SDS: After Dose 1 (N=250) | 13vPnC MDV: After Dose 2 (N=249) | 13vPnC SDS: After Dose 2 (N=248) | 13vPnC MDV: After Dose 3 (N=247) | 13vPnC SDS: After Dose 3 (N=244) | Screened Only (N=26)
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 3 | 3 | 3 | 1 | 4 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 27 | 17 | 17 | 10 | 19 | 25 | 0
Viral diarrhoea (Infections and infestations) | 0 | 0 | 6 | 10 | 8 | 10 | 5 | 10 | 0
Tinea capitis (Infections and infestations) | 0 | 0 | 4 | 3 | 3 | 1 | 2 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 3 | 1 | 1 | 3 | 0 | 4 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 2 | 2 | 1 | 3 | 2 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 (0)
Dysentery (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Injection site abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 3 | 6 | 3 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinea faciei (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 (0)
Chest wall abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 8 | 12 | 5 | 7 | 2 | 6 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Vaccination site swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Redness: Any (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 1/248 | 0 | 2/247 | 0/247 | 0/246 | 0/241 | 0
Redness: Mild (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 1/248 | 0 | 2/247 | 0/247 | 0/246 | 0/241 | 0
Redness: Moderate (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/248 | 0 | 0/247 | 0/247 | 0/246 | 0/241 | 0
Redness: Severe (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/248 | 0 | 0/247 | 0/247 | 0/246 | 0/241 | 0
Swelling: Any (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 1/248 | 0 | 2/247 | 0/247 | 0/246 | 0/241 | 0
Swelling: Mild (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 1/248 | 0 | 2/247 | 0/247 | 0/246 | 0/241 | 0
Swelling: Moderate (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/248 | 0 | 1/247 | 0/247 | 0/246 | 0/241 | 0
Swelling: Severe (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/248 | 0 | 0/247 | 0/247 | 0/246 | 0/241 | 0
Tenderness: Any (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 42/248 | 47 | 34/248 | 32/247 | 37/246 | 35/241 | 0
Tenderness: Mild (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 32/248 | 37 | 27/248 | 28/247 | 30/246 | 32/241 | 0
Tenderness: Moderate (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 13/248 | 14 | 7/247 | 5/247 | 9/246 | 4/241 | 0
Tenderness: Severe (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/248 | 0 | 0/247 | 0/247 | 0/246 | 0/241 | 0
Fever: >=38.0 degree C (General disorders) | 0/0 | 0/0 | 9/248 | 7 | 7/247 | 7/247 | 3/246 | 8/241 | 0
Fever: >=38.0 but <=39.0 degrees C (General disorders) | 0/0 | 0/0 | 9/248 | 7 | 7/247 | 7/247 | 3/246 | 7/241 | 0
Fever: >39.0 but <=40.0 degrees C (General disorders) | 0/0 | 0/0 | 0/248 | 0 | 1/247 | 0/247 | 0/246 | 1/241 | 0
Fever: >40.0 degrees C (General disorders) | 0/0 | 0/0 | 0/248 | 0 | 0/247 | 0/247 | 0/246 | 0/241 | 0
Decreased appetite: Any (General disorders) | 0/0 | 0/0 | 17/248 | 26 | 28/247 | 18/247 | 24/246 | 20/242 | 0
Decreased appetite: Moderate (General disorders) | 0/0 | 0/0 | 17/248 | 26 | 28/247 | 18/247 | 24/246 | 19/242 | 0
Decreased appetite: Severe (General disorders) | 0/0 | 0/0 | 0/248 | 0 | 0/247 | 0/247 | 0/246 | 1/241 | 0
Irritability: Any (General disorders) | 0/0 | 0/0 | 103/249 | 93 | 93/248 | 83/247 | 83/246 | 92/243 | 0
Irritability: Mild (General disorders) | 0/0 | 0/0 | 86/249 | 77 | 75/248 | 67/247 | 71/246 | 74/242 | 0
Irritability: Moderate (General disorders) | 0/0 | 0/0 | 19/248 | 17 | 23/247 | 17/247 | 15/246 | 18/242 | 0
Irritability: Severe (General disorders) | 0/0 | 0/0 | 0/248 | 0 | 0/247 | 3/247 | 1/246 | 5/241 | 0
Increased sleep: Any (General disorders) | 0/0 | 0/0 | 16/248 | 14 | 24/247 | 14/247 | 12/246 | 12/241 | 0
Increased sleep: Mild (General disorders) | 0/0 | 0/0 | 11/248 | 10 | 20/247 | 12/247 | 10/246 | 11/241 | 0
Increased sleep: Moderate (General disorders) | 0/0 | 0/0 | 6/248 | 4 | 4/247 | 1/247 | 2/246 | 1/241 | 0
Increased sleep: Severe (General disorders) | 0/0 | 0/0 | 0/248 | 0 | 0/247 | 1/247 | 1/246 | 0/241 | 0
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Growth retardation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.